CLINICAL TRIAL: NCT01771367
Title: A Clinical Study to Generate an Exploratory Training Set of Data Characterising Clinical Events, Physiological and Metabolic Responses, and Innate and Adaptive Immune Responses Following a Single Intramuscular Immunisation With Either "Fluad" or "Agrippal" Influenza Vaccines or Saline Placebo in Healthy Adults.
Brief Title: Training Study to Characterize Biomarkers to Flu Vaccines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CRC305C
Record Dates: First submitted 2013-01-15; First posted 2013-01-18 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
MeSH Terms: interventions — fluad vaccine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluad (Active Comparator): Participants receive one dose of Fluad vaccine.
  Interventions: Biological: Fluad
- Agrippal (Active Comparator): Participants receive one dose of Agrippal vaccine.
  Interventions: Biological: Agrippal
- Placebo (Placebo Comparator): Participants receive one dose of saline placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Fluad
  Arms: Fluad
Biological: Agrippal
  Arms: Agrippal
Biological: Placebo
  Arms: Placebo

SUMMARY:
It is thought that vaccines trigger innate inflammatory responses to induce antigen-specific adaptive immunity (the desired effect), but excessive inflammation may lead to serious inflammatory complications or unwanted side effects. Currently there is a lack of reliable biomarkers (a measurable biological response that predicts something) able to predict severe inflammation and this has resulted in the development of several vaccines being terminated and the withdrawal of some licensed vaccines which were associated with inflammatory complications.

This study is part of the BIOVACSAFE project which is a 5-year 30 million Euro project funded by the Innovative Medicines Initiative. The project involves a series of clinical studies using licensed vaccines as benchmarks to generate clinical data on inflammation and identify biomarkers that can be used to predict acceptable reactogenicity. The target is to identify biomarkers that can predict the occurrence of beneficial and detrimental effects in response to a vaccine. Such biomarkers could be used in future vaccine development programs to optimise selection of vaccine candidates with a profile that will be unlikely to generate worrisome safety signals once they are in generalised use.

This study is one in a series of "training" studies which will each use different licensed vaccines that are prototypical representatives of a class of vaccine used in a particular population. Forty-eight subjects will be randomised into three groups to receive: a) Fluad (n=20), b) Agrippal (n=20), c) saline placebo (n=8). Following a screening visit, participants will undergo a seven-day residential visit which will include immunisation and intensive monitoring of physiological (e.g. heart rate, oral temperature, blood pressure) metabolic and immune (innate and adaptive) parameters. This visit will be followed up by four outpatient visits with further monitoring and blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged 18-45 years inclusive. Randomisation will ensure equal numbers of men and women.
2. The subject is, in the opinion of the investigator, healthy on the basis of medical history, vital signs, and the results of routine laboratory tests with no active disease process that could interfere with the study endpoints.
3. Body Mass Index ≥18.5 and <29.5
4. The subject is able to read and understand the Informed Consent Form (ICF), and understand study procedures.
5. The subject has signed the ICF.
6. Available for follow-up for the duration of the study.
7. Agree to abstain from donating blood during and for three months after the end of their participation in the study, or longer if necessary.
8. If heterosexually active female, willing to use an effective method of contraception with partner (oral contraceptive pill; intrauterine device; injectable or implanted contraceptive; condoms incorporating spermicide if using these; physiological or anatomical sterility) from 30 days prior to, and 3 months after, vaccination. Willing to undergo urine pregnancy tests prior to vaccination and blood pregnancy test at screening and final follow up.
9. The subject self-reports at screening that for the past month they have had regular sleep pattern with bedtime occurring between 22:00 and 01:00 h.
10. The subject has venous access sufficient to allow blood sampling as per the protocol.

Exclusion Criteria:

1. Significant dietary restrictions (e.g. vegan, lactose intolerant, but vegetarian acceptable) or life-threatening food allergies (e.g. anaphylaxis-related nut allergies).
2. Pregnant or lactating at any point during the study from screening to final follow up.
3. As subjects must be eligible to be randomised to any of the treatment groups they must fulfil the vaccine contraindications eligibility for both group A & B:

   1. Hypersensitivity to the active components of FLUAD, any of the excipients, eggs, chicken proteins, kanamycin and neomycin sulphate, formaldehyde, and cetyltrimetholammonium bromide or those who have had a previous life-threatening reaction to previous influenza vaccinations.
   2. Hypersensitivity to the active substances of Agrippal, to any excipients and to residues such as eggs and chicken proteins including ovalbumin.
4. Presence of primary or acquired immunodeficiency states with a total lymphocyte count less than 1,200 per mm3 or presenting other evidence of lack of cellular immune competence e.g. leukaemias, lymphomas, blood dyscrasias, or patients receiving immunosuppressive therapy (including regular use of oral, inhaled, topical or parenteral corticosteroids).
5. Use of any immune suppressing or immunomodulating drugs within 6 months of Visit 1 (screening).
6. Regular use of non-steroidal anti-inflammatory drugs (by any route of administration including topical) within 6 months of Visit 1 (screening) considered by the study physician as likely to interfere with immune responses.
7. Receipt of a vaccine within 30 days of visit 2, or requirement to receive another vaccine within the study period.
8. Presence of an acute severe febrile illness at time of immunisation.
9. History of alcohol, narcotic, benzodiazepine, or other substance abuse or dependence within the 12 months preceding Visit 1.
10. Currently participating in another clinical study with an investigational or non-investigational drug or device, or has participated in a clinical trial within the 3 months preceding Visit 1.
11. Any condition that, in the investigator's opinion, compromises the subject's ability to meet protocol requirements or to complete the study.
12. Receipt of blood products or immunoglobin, or blood donation, within 3 months of screening.
13. Unable to read and speak English to a fluency level adequate for the full comprehension of procedures required in participation and consent.
14. An average weekly alcohol intake that exceeds 14 or 21 units per week for females and males, respectively (1 unit = 12 oz or 360ml of beer; 5oz or 150ml of wine; 1.5oz or 45ml of distilled spirits), or unwilling to stop alcohol consumption for each treatment period during the study.
15. Currently smokes in excess of 5 cigarettes/day or use tobacco or nicotine substitutes (within the last 6 months of screening), or subjects unwilling to refrain from smoking or are unable to abide by Surrey CRC restrictions.
16. Consumes excessive amounts, defined as greater than 4 servings (1 serving is approximately equivalent to 120mg caffeine) of coffee, tea, cola, or other caffeinated beverages/food per day.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline values of global gene expression in whole blood. | Visits 1 (Day -28 to -2), 2 (Day -1 to +5) , 3 (Day 7), 4 (Day 14), 5 (Day 21), 6 (Day 28).

OTHER OUTCOMES:
Proportion of subjects experiencing vaccine-related clinical events following administration of first dose of vaccine. | Visits 2 (Day -1 to +5) , 3 (Day 7), 4 (Day 14), 5 (Day 21) and 6 (Day 28).

CONTACTS AND LOCATIONS:
Overall Officials: David Lewis, Principal Investigator — University of Surrey
Locations (1):
- University of Surrey, (Surrey Clinical Research Centre), Guildford, Surrey, United Kingdom

REFERENCES:
- [Derived] Weiner J, Lewis DJM, Maertzdorf J, Mollenkopf HJ, Bodinham C, Pizzoferro K, Linley C, Greenwood A, Mantovani A, Bottazzi B, Denoel P, Leroux-Roels G, Kester KE, Jonsdottir I, van den Berg R, Kaufmann SHE, Del Giudice G. Characterization of potential biomarkers of reactogenicity of licensed antiviral vaccines: randomized controlled clinical trials conducted by the BIOVACSAFE consortium. Sci Rep. 2019 Dec 30;9(1):20362. doi: 10.1038/s41598-019-56994-8. PMID 31889148
- [Derived] Muturi-Kioi V, Lewis D, Launay O, Leroux-Roels G, Anemona A, Loulergue P, Bodinham CL, Aerssens A, Groth N, Saul A, Podda A. Neutropenia as an Adverse Event following Vaccination: Results from Randomized Clinical Trials in Healthy Adults and Systematic Review. PLoS One. 2016 Aug 4;11(8):e0157385. doi: 10.1371/journal.pone.0157385. eCollection 2016. PMID 27490698
- [Derived] Spensieri F, Siena E, Borgogni E, Zedda L, Cantisani R, Chiappini N, Schiavetti F, Rosa D, Castellino F, Montomoli E, Bodinham CL, Lewis DJ, Medini D, Bertholet S, Del Giudice G. Early Rise of Blood T Follicular Helper Cell Subsets and Baseline Immunity as Predictors of Persisting Late Functional Antibody Responses to Vaccination in Humans. PLoS One. 2016 Jun 23;11(6):e0157066. doi: 10.1371/journal.pone.0157066. eCollection 2016. PMID 27336786
- See also: BIOVACSAFE — http://www.biovacsafe.eu/